CLINICAL TRIAL: NCT06755476
Title: The Effect of Psychological Counseling Program (PsychoCP) for Alzheimer's Patients' Caregivers on Perceived Stress, Psychological Well-Being and Caregiver Burden
Brief Title: Psychological Counseling Program for Alzheimer's Patients' Caregivers
Acronym: PsychoCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydan Akkurt Yalçıntürk (Other)
Responsible Party: Sponsor-Investigator, Aydan Akkurt Yalçıntürk, Asst. Prof., Uskudar University
Organization: Uskudar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20122024
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease; Caregivers of Alzheimer's Disease or Memory Problem Patients; Perceived Stress; Well-Being (Psychological Flourishing); Care Burden
MeSH Terms: conditions — Alzheimer Disease; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PsychoCP (Experimental)
  Interventions: Other: Psychological Counseling Program
- Control (No Intervention)

INTERVENTIONS:
Other: Psychological Counseling Program — The Psychological Counseling Program consists of 8 sessions for caregivers of individuals diagnosed with Alzheimer's.
  Aims of the sessions:
  Session 1: Introduction, Collection of pretest data Session 2: It is aimed to inform Alzheimer's caregivers about the disease and its symptoms.
  Session 3: It is aimed to strengthen caregivers' coping skills. Session 4: It is aimed to inform Alzheimer's patients about daily care practices.
  Session 5: It is aimed to provide information to Alzheimer's caregivers about coping with stress.
  Session 6: It is aimed to provide information about medical and financial support that individuals diagnosed with Alzheimer's and their relatives can receive in the region they live.
  Session 7: It is aimed to conduct Q&A sessions on the problems that caregivers bring.
  Session 8: Collection of posttest data Sessions will be completed in 8 weeks, one day a week. Each session is planned to last approximately 60 minutes.
  Arms: PsychoCP

SUMMARY:
Purpose: To investigate the effects of a psychological counseling program (PsychoCP) applied to caregivers of Alzheimer's patients on perceived stress, psychological well-being and care burden.

Design: The study will be conducted in a pre-test post-test control group, randomized controlled experimental research design.

Method: The study is planned to be carried out in Bağcılar Municipality Vefahâne Life Center, Antalya Alzheimer Patients and Patient Relatives Meeting Center and Osmaniye Family and Social Policies Directorate. The sample of the study will consist of 80 caregivers. They will be assigned to intervention (n=40) and control groups (n=40) by randomization.

Hypotheses Hypothesis1: The perceived stress level of caregivers who received PsychoDP is lower than those who did not receive PsychoCP.

Hypothesis2: The psychological well-being levels of caregivers who received PsychoDP are higher than those who did not receive PsychoCP.

Hypothesis3: The care burden of caregivers who received PsychoDP is lower than those who did not receive PsychoCP.

ELIGIBILITY:
Inclusion Criteria:

* Providing informal care to an individual with mild or moderate Alzheimer's disease
* Being a primary caregiver
* Providing care to the patient for at least six months
* Providing care to the patient for at least six hours per day
* Being literate
* Being able to speak and understand Turkish
* Being 18 years of age or older
* Being willing and able to participate in the study

Exclusion Criteria:

* Not being able to understand questions and express ideas
* Having a psychiatric disorder
* Not receiving any therapy services during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Level | Two months
  Perceived Stress Scale: It was developed to measure the stress level of specific situations in individuals' lives. This scale consists of 14 items and is evaluated by participants on a 5-point Likert-type scale ranging from "never (0)" to "very often (4)". The score range of the scale is 0-56. High scores obtained from the scale indicate that the individual's perceived stress level is high.
Psychological Well-being Level | Two months
  Psychological Well-being Scale: It is a scale that evaluates the psychological well-being of an individual. The items of the scale are rated between 1 and 7 as strongly disagree (1) and strongly agree (7). The minimum score is 8 and the maximum score is 56. An increase in the score value indicates that the person has many psychological resources and strengths.
The Burden of Caregiving | Two months
  Zarit Caregiver Burden Scale: The scale is used to measure the stress of caregivers. It contains 22 Likert-type statements. The statements range from zero to four as never (0), rarely (1), sometimes (2), quite often (3), almost always (4). A minimum of 0 and a maximum of 88 points can be obtained from the scale. As the score value increases, the stress experienced by the caregiver also increases.

IPD SHARING:
Plan to Share IPD: No